CLINICAL TRIAL: NCT02344602
Title: A Deep Phenotyping Approach to Assess the Effect of Uric Acid Lowering in Patients With Uncomplicated Type 1 Diabetes Mellitus
Brief Title: The Effect of Uric Acid Lowering in Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Toronto General Hospital (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, David Z.I. Cherney, MD, PhD, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-5427-A
Record Dates: First submitted 2015-01-09; First posted 2015-01-26 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetic Nephropathy; Diabetes Mellitus; Diabetes Complications; Uric Acid; Febuxostat; Uloric; Glomerular Filtration Rate; Kidney Disease; Vascular Disease; Cardiovascular Diseases; Endothelial Function; Arterial Stiffness; Pharmacologic Actions; Gout Suppressants; Therapeutic Uses; Free Radical Scavengers; Antioxidants; Protective Agents; Physiological Effects of Drugs; Angiotensin II Infusion; Flow-mediated Dilation; Flow-mediated Constriction; Nitroglycerin; Hyperglycemia; Renin-angiotensin-aldosterone System; Nitric Oxide; cGMP; Oxidative Stress; Renal Haemodynamic Function; Inulin Clearance; PAH Clearance; Skin Biopsy; T1R mRNA Expression; Cytokines; Chemokines
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies; Diabetes Mellitus; Diabetes Complications; Kidney Diseases; Vascular Diseases; Cardiovascular Diseases; Hyperglycemia | interventions — Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Febuxostat (trade name Uloric®) (Experimental): Oral tablet, 80mg, OD, 8 weeks
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Febuxostat — Oral tablet, 80mg, OD, 8 weeks
  Other Names: Trade name Uloric®

SUMMARY:
Patients with type 1 diabetes mellitus (T1DM) are at high risk of developing kidney complications potentially leading to end stage renal disease. Uric acid (UA), the end product of purine metabolism, emerged as an important determinant of renal and vascular injury due to its ability activate the renin-angiotensin-aldosterone system (RAAS) and increase production of harmful reactive oxygen species (ROS). ROS cause progressive endothelial cell dysfunction, inflammation, tissue fibrosis and eventually cell death. These processes are enhanced in DM because of the effect of hyperglycemia.

Since existing preventive drug therapies fail to completely prevent kidney damage, an examination of the effect of UA lowering against initiation and progression of renal and vascular complications is therefore of the utmost importance. The purpose of this study is to examine the effect of UA lowering with febuxostat on renal and systemic vascular function in patients with uncomplicated T1DM. It was hypothesized that UA lowering will improve kidney and systemic vascular function through effects on blood vessel function and anti-inflammatory effect.

Kidney and blood vessel function will be assessed under conditions of normal and high blood sugar levels before and after 8 weeks of treatment with the UA lowering drug febuxostat in patients with diabetes and during normoglycemia only in health controls.

Current treatment for renal and vascular complications in DM patients includes blockade of the RAAS. Unfortunately, angiotensin converting enzyme inhibitors (ACEi) and angiotensin II (AngII) receptor blockers (ARBs) lead to incomplete RAAS suppression, and do not completely prevent renal or vascular complications. Moreover, dual RAAS blockade increases renal and cardiovascular risk. Recent experimental work suggests that UA lowering therapies can block the RAAS, suppress inflammation and promote renal and systemic vascular protection. Therefore, our study is critical in determining the possible role of early UA lowering on renal and systemic hemodynamic dysfunction in young patients with T1DM.

DETAILED DESCRIPTION:
Uric acid (UA) was recently suggested to exert deleterious effects on blood pressure and renal function, even when baseline UA levels are within the normal range. UA activates the renin angiotensin-aldosterone system (RAAS), increases oxidative stress and promotes inflammation. As a consequence, higher UA levels are associated with metabolic abnormalities (insulin resistance, hyperglycemia), cardiovascular disease (hypertension, endothelial dysfunction, arterial stiffness, cardiac diastolic dysfunction) and kidney function abnormalities (hyperfiltration - a marker for intraglomerular hypertension, proteinuria). Thus pharmacologic UA lowering may promote renal and cardiovascular protection. The mechanisms underlying these protective effects in humans, prior to the onset of clinical disease, remain unknown.

This study is focused on the prevention of complications in young, normotensive type 1 diabetes mellitus (T1DM) patients with normal renal function and UA levels. The study will examine the effect of UA lowering with febuxostat (FBX) on renal hemodynamic function, vascular function and urinary inflammatory biomarkers. Based on substantial supportive pre-clinical and epidemiological data, we hypothesize that lowering UA levels that are within normal range at baseline will: 1) ameliorate hemodynamic abnormalities characteristic of T1DM, and reduce renal and systemic hypertensive responses to hyperglycemia; 2) ameliorate endothelial function abnormalities characteristic of T1DM; 3) reduce urinary inflammatory cytokines/chemokine excretion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years old
* Normoalbuminuria 24 hour urine collection
* Body mass index 18-30 kg/m2 at screening
* Subject able, willing to perform assessments
* Normal electrocardiogram
* Normal renal (estimated GFR>60 ml/min)
* Clinic blood pressure <140/90 mmHg
* Type 1 DM, duration of diabetes >1 years
* Able to take medications every day
* Signed and dated written informed consent on the screening visit in accordance with GCP and local legislation
* Hemoglobin A1c 6-11%
* Normal uric acid levels

Exclusion Criteria:

* Cardiac, lung or peripheral vascular disease or stroke, gout
* Hypertension, or on BP-lowering medicine
* History of proliferative retinopathy
* Diagnosis of brittle diabetes based on investigator judgement
* Allergy to either allopurinol or probenecid
* Pregnancy, breastfeeding, no reliable contraception
* Oral contraceptives (due to effects on the RAS)
* Alcohol or tobacco within 24 hours prior to the study
* Uric acid ≥420 μmol/L or taking uric acid lowering agents
* Use of agents that influence GFR or interfere with purine metabolism (didanosine, azothioprine, methotrexate, NSAIDs, mycophenolate)
* Pancreas, pancreatic islet cells or renal transplant recipient
* Medical history of cancer or treatment for cancer in the last five years prior to screening
* T1DM treatment with any other drugs to reduce blood glucose except insulin within 6 months prior to screening (example: off-label use of metformin)
* Known autonomic neuropathy and proliferative retinopathy including treated proliferative retinopathy. Subjects with mild non-proliferative diabetic retinopathy can be included
* Alcohol or drug abuse within the three months prior to informed consent that would interfere with trial participation based on investigator judgement or any ongoing clinical condition that would jeopardize subject safety or study compliance based on investigator judgement
* ACE inhibitors, angiotensin receptor blockers, direct renin inhibitors, aldosterone antagonists
* Indication of liver disease, defined by serum levels of either alanine transaminase (ALT) (SGPT), aspartate transaminase (AST) (SGOT), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined during screening
* Blood disorders causing hemolysis or unstable red blood cells (e.g. malaria, hemolytic anemia)
* Pre-menopausal women (last menstruation ≤ 1 year prior to informed consent) who are nursing or pregnant or are of child-bearing potential and are not practising an acceptable method of birth control, or do not plan to continue using this method throughout the study.
* Participation in another trial with an investigational drug within 30 days prior to informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2012-12-18 (Actual); Primary Completion 2015-09-22 (Actual); Study Completion 2015-09-22 (Actual)

PRIMARY OUTCOMES:
The Change in Glomerular Filtration Rate (GFR) After an 8 week Treatment with Febuxostat | Before and after an 8 week treatment with febuxostat.
  Glomerular filtration rate (GFR, based on inulin plasma clearance) will be measured in euglycemic and hyperglycemic conditions before and after an 8 week treatment with febuxostat and in response to 1 ng/kg/min and 3 ng/kg/min Angiotensin II infusions in euglycemic conditions before and after 8 weeks of febuxostat administration.
The Change in Effective Renal Plasma Flow (ERPF) After an 8 week Treatment with Febuxostat | Before and after an 8 week treatment with febuxostat
  Effective Renal Plasma Flow (ERPF, based on paraaminohippurate plasma clearance) will be measured in euglycemic and hyperglycemic conditions before and after an 8 week treatment with febuxostat and in response to 1 ng/kg/min and 3 ng/kg/min Angiotensin II infusions in euglycemic conditions before and after 8 weeks of febuxostat administration.

SECONDARY OUTCOMES:
The Change in Renin Angiotensin Aldosterone System (RAAS) Markers and Neurohormonal Activation After an 8 week Treatment with Febuxostat | Before and after an 8 week treatment with febuxostat.
  RAAS and neurohormonal markers will be measured in euglycemic and hyperglycemic conditions before and after an 8 week treatment with febuxostat.
The Change in Levels of Vasodilators in Plasma After an 8 week Treatment with Febuxostat | Before and after an 8 week treatment with febuxostat.
  Levels of vasodilators will be measured in plasma in euglycemic and hyperglycemic conditions before and after an 8 week treatment with febuxostat.
The Change in Blood Pressure After an 8 week Treatment with Febuxostat | Before and after an 8 week treatment with febuxostat.
  Blood pressure in euglycemic and hyperglycemic conditions before and after an 8 week treatment with febuxostat and in response to 1 ng/kg/min and 3 ng/kg/min Angiotensin II infusions in euglycemic conditions before and after 8 weeks of febuxostat administration.
The Change in Flow Mediated Dilation After an 8 week Treatment with Febuxostat | Before and after an 8 week treatment with febuxostat.
  Flow Mediated Dilation will be measured in euglycemic and hyperglycemic conditions before and after an 8 week treatment with febuxostat.
The Change in Arterial Stiffness After an 8 week Treatment with Febuxostat | Before and after an 8 week treatment with febuxostat.
  Arterial Stiffness will be measured in euglycemic and hyperglycemic conditions before and after an 8 week treatment with febuxostat.
The Change in Skin Biopsy Measures of Neurohormonal Activation After an 8 week Treatment with Febuxostat | Before and after an 8 week treatment with febuxostat.
  Skin biopsy neurohormonal activation biomarkers will be measured in euglycemic conditions before and after an 8 week treatment with febuxostat.

CONTACTS AND LOCATIONS:
Overall Officials: David ZI Cherney, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Renal Physiology Laboratory, University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lytvyn Y, Har R, Locke A, Lai V, Fong D, Advani A, Perkins BA, Cherney DZI. Renal and Vascular Effects of Uric Acid Lowering in Normouricemic Patients With Uncomplicated Type 1 Diabetes. Diabetes. 2017 Jul;66(7):1939-1949. doi: 10.2337/db17-0168. Epub 2017 Apr 13. PMID 28408434